CLINICAL TRIAL: NCT01620034
Title: A Randomized Study of Stereotactic Body Radiotherapy (SBRT) for Lung Tumours Delivered Over 4 Days Versus 11 Days
Brief Title: Lung Stereotactic Body Radiotherapy (SBRT) Delivered Over 4 Days Versus 11 Days
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Patrick Cheung, Radiation Oncologist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 106-2010
Record Dates: First submitted 2012-06-11; First posted 2012-06-15 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Peripherally Located Stage I Lung Cancer; Peripherally Located Solitary Lung Metastasis
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 11 Day Arm (Active Comparator)
  Interventions: Radiation: Stereotactic Body Radiotherapy
- 4 Day Arm (Experimental)
  Interventions: Radiation: Stereotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy — Patients on the 11 day arm receive 4 fractions of SBRT every 3rd day. Patients on the 4 day arm receive 4 fractions of SBRT every day.

SUMMARY:
Stereotactic Body Radiotherapy (SBRT) has emerged as a new treatment option for peripherally located lung tumours, offering very high rates of tumour eradication, with minimal side effects. Even though this treatment option is being adopted in more and more cancer centres, there is still no consensus about the optimal schedule for the radiation treatment. Generally speaking, most lung SBRT schedules involve delivering 3-4 days of radiation. At the Sunnybrook Odette Cancer Centre, the lung SBRT policy is to deliver 4 days of radiation over 11 days (each treatment given once very 3rd day). However, some centres deliver the same treatment over 4 days in a row (each treatment given once daily over 4 days). There is no evidence from the published literature to suggest that there is any difference in side effects between delivering the SBRT over 4 days versus 11 days. To confirm this, the investigators propose to conduct a comparative (randomized) study to compare these 2 approaches.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of malignancy in the lung (either NSCLC or metastasis)
* If pathologic diagnosis is not available, there must be evidence of FDG uptake on PET-CT suggestive of malignancy and/or evidence of tumour growth over serial CT scans
* Clinical stage I lung cancer or solitary lung metastasis located in the periphery away from central mediastinal structures and <=5cm in size
* Patient deemed suitable for lung SBRT (reasonable performance status, acceptable pulmonary function) by the attending Radiation Oncologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Rate of grade 2 or higher acute toxicity | Within 4 months after completion of therapy
  CTCAE v4.0 will be used to capture radiotherapy toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Cheung, MD, FRCPC, Principal Investigator — Toronto Sunnybrook Regional Cancer Centre
Locations (1):
- Sunnybrook Odette Cancer Centre, Toronto, Ontario, Canada